CLINICAL TRIAL: NCT02706847
Title: A Phase 3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) to Placebo on Stable Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs) in Subjects With Moderately to Severely Active Rheumatoid Arthritis With Inadequate Response or Intolerance to Biologic DMARDs (bDMARDs)
Brief Title: A Study to Compare Upadacitinib (ABT-494) to Placebo in Adults With Rheumatoid Arthritis on Stable Dose of Conventional Synthetic Disease-Modifying Antirheumatic Drugs (csDMARDs) With an Inadequate Response or Intolerance to Biologic DMARDs
Acronym: SELECT-BEYOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-542; 2015-003335-35 (EudraCT Number)
Record Dates: First submitted 2016-02-18; First posted 2016-03-11 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Musculoskeletal Disease; Arthritis; Joint Disease; Anti-inflammatory agents; Antirheumatic agents; ABT-494; upadacitinib
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Upadacitinib 15 mg (Experimental): Period 1: Participants receive upadacitinib 15 mg once daily for 24 weeks.
  Period 2: Participants will continue on upadacitinib 15 mg once daily from Week 24 to Week 260.
  Interventions: Drug: Upadacitinib
- Upadacitinib 30 mg (Experimental): Period 1: Participants receive upadacitinib 30 mg once daily for 24 weeks.
  Period 2: Participants continue on upadacitinib 30 mg once daily until implementation of Protocol Amendment 4, then participants begin to receive upadacitinib 15 mg once daily up to Week 260.
  Interventions: Drug: Upadacitinib
- Placebo / Upadacitnib 15 mg (Placebo Comparator): Period 1: Participants receive placebo once daily for 12 weeks followed by upadacitinib 15 mg once daily for 12 weeks.
  Period 2: Participants will continue on upadacitinib 15 mg once daily from Week 24 to Week 260.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- Placebo / Upadacitnib 30 mg (Placebo Comparator): Period 1: Participants receive placebo once daily for 12 weeks followed by upadacitinib 30 mg once daily for 12 weeks.
  Period 2: Participants continue on upadacitinib 30 mg once daily until implementation of Protocol Amendment 4, then participants begin to receive upadacitinib 15 mg once daily up to Week 260.
  Interventions: Drug: Placebo; Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Tablet; Oral
  Arms: Placebo / Upadacitnib 15 mg; Placebo / Upadacitnib 30 mg
Drug: Upadacitinib — Tablet; Oral
  Other Names: ABT-494; RINVOQ®

SUMMARY:
The study objective of Period 1 (Day 1 to Week 24) is to compare the safety and efficacy of upadacitinib 30 mg once daily (QD) and 15 mg QD versus placebo for the treatment of signs and symptoms of participants with moderately to severely active rheumatoid arthritis (RA) who are on a stable dose of csDMARDs and had an inadequate response to or intolerance to at least 1 bDMARD.

The study objective of Period 2 (Week 24 to Week 260) is to evaluate the long-term safety, tolerability, and efficacy of upadacitinib 15 mg QD and 30 mg QD in participants with RA who completed Period 1.

DETAILED DESCRIPTION:
This study includes a 35-day screening period; a 24-week randomized, double-blind, parallel-group, placebo controlled treatment period (Period 1); a 236-week blinded long-term extension period (Period 2); and a 30-day follow-up period (call or visit).

Period 1 consists of a 12-week double-blind, placebo-controlled treatment phase plus a 12-week double-blind phase where all participants were to receive upadacitinib; at Week 12 participants assigned to placebo will be switched to upadacitinib according to their randomization assignment.

Participants who meet eligibility criteria will be randomized in a 2:2:1:1 ratio to one of four treatment groups:

* Group 1: Upadacitinib 30 mg QD (Day 1 to Week 12) → upadacitinib 30 mg QD (Week 12 and thereafter)
* Group 2: Upadacitinib 15 mg QD (Day 1 to Week 12) → upadacitinib 15 mg QD (Week 12 and thereafter)
* Group 3: Placebo (Day 1 to Week 12) → upadacitinib 30 mg QD (Week 12 and thereafter)
* Group 4: Placebo (Day 1 to Week 12) → upadacitinib 15 mg QD (Week 12 and thereafter)

Participants will continue stable dose of csDMARD therapy for the first 24 weeks of the study.

Participants who complete the Week 24 visit (end of Period 1) will enter the blinded long-term extension portion of the study, Period 2 and continue to receive the same dose of upadacitinib per original randomization assignment in a blinded manner. Starting at Week 24, at least 20% improvement in both swollen joint count (SJC) and tender joint count (TJC) compared to Baseline is required to remain on study drug. Starting at Week 24, initiation of or change in corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, or adding or increasing doses in up to 2 csDMARDs (concomitant use of up to 2 csDMARDs except the combination of methotrexate and leflunomide) is allowed as per local label.

With the implementation of Protocol Amendment 4, all participants in the extension period will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) for≥ 3 months.
* Treated for ≥ 3 months with ≥ 1 bDMARD therapy, but continue to exhibit active RA or had to discontinue due to intolerability or toxicity, irrespective of treatment duration prior to the first dose of study drug.
* Participant has been receiving csDMARD therapy ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug. The following csDMARDs are allowed: methotrexate (MTX), sulfasalazine, hydroxychloroquine, chloroquine, and leflunomide. A combination of up to two background csDMARDs is allowed except the combination of MTX and leflunomide.
* Meets both of the following criteria:
* ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits.
* hsCRP ≥ 3mg/L at Screening Visit.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than RA (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial spondyloarthritis, reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, fibromyalgia [currently with active symptoms]). Current diagnosis of secondary Sjogren's Syndrome is permitted.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (188):
- United States (103):
  - Rheum Assoc of North Alabama /ID# 145959, Huntsville, Alabama
  - AZ Arthritis and Rheum Assoc /ID# 148593, Mesa, Arizona
  - AZ Arthritis and Rheum Researc /ID# 142816, Phoenix, Arizona
  - AZ Arthritis and Rheum Researc /ID# 146075, Phoenix, Arizona
  - AZ Arthritis and Rheum Researc /ID# 148592, Phoenix, Arizona
  - Arizona Research Center, Inc. /ID# 142741, Phoenix, Arizona
  - AZ Arthr & Rheum Research /ID# 155256, Prescott, Arizona
  - AZ Arthritis & Rheum Research /ID# 156090, Sun City, Arizona
  - NEA Baptist Clinic /ID# 149280, Jonesboro, Arkansas
  - Covina Arthritis Clinic /ID# 142794, Covina, California
  - Rheumatology Ctr of San Diego /ID# 153576, Escondido, California
  - St. Joseph Heritage Healthcare /ID# 149273, Fullerton, California
  - TriWest Research Associates- La Mesa /ID# 142792, La Mesa, California
  - Arthritis & Osteo Medical Ctr /ID# 142770, La Palma, California
  - Valerius Med Grp & Res Ctr /ID# 142799, Los Alamitos, California
  - Pacific Arthritis Ctr Med Grp /ID# 142783, Los Angeles, California
  - University of California, Los Angeles /ID# 148348, Los Angeles, California
  - Desert Medical Advances /ID# 142765, Palm Desert, California
  - Stanford University School of Med /ID# 142761, Stanford, California
  - Robin K. Dore MD, Inc /ID# 150908, Tustin, California
  - Inland Rheum Clin Trials Inc. /ID# 142787, Upland, California
  - Medvin Clinical Research /ID# 142814, Whittier, California
  - Arthritis Assoc & Osteo Ctr /ID# 142809, Colorado Springs, Colorado
  - Denver Arthritis Clinic /ID# 142771, Denver, Colorado
  - New England Research Associates, LLC /ID# 142763, Bridgeport, Connecticut
  - Delaware Arthritis /ID# 142803, Lewes, Delaware
  - Lakes Research, LLC /ID# 142755, Miami, Florida
  - Medallion Clinical Research Institute, LLC /ID# 142740, Naples, Florida
  - Omega Research Consultants /ID# 142780, Orlando, Florida
  - Millennium Research /ID# 142782, Ormond Beach, Florida
  - Arthritis Research of Florida /ID# 142811, Palm Harbor, Florida
  - Arthritis Center, Inc. /ID# 142822, Palm Harbor, Florida
  - Advent Clinical Research /ID# 142817, Pinellas Park, Florida
  - St. Anthony Comprehsve Res Ins /ID# 148349, St. Petersburg, Florida
  - University of South Florida /ID# 145611, Tampa, Florida
  - BayCare Medical Group, Inc. /ID# 142747, Tampa, Florida
  - Lovelace Scientific Resources /ID# 142779, Venice, Florida
  - Jefrey D. Lieberman, MD, P.C. /ID# 151713, Decatur, Georgia
  - Marietta Rheumatology Assoc /ID# 151347, Marietta, Georgia
  - St. Luke's Clinic - Rheumatolo /ID# 150923, Boise, Idaho
  - Institute of Arthritis Res /ID# 142810, Idaho Falls, Idaho
  - Advanced Clinical Research /ID# 153089, Meridian, Idaho
  - Great Lakes Clinical Trials /ID# 148341, Chicago, Illinois
  - Clinical Investigation Special /ID# 149270, Skokie, Illinois
  - Springfield Clinic /ID# 142818, Springfield, Illinois
  - Deerbrook Medical Associates /ID# 151712, Vernon Hills, Illinois
  - The Arthritis & Diabetes Clinic, Inc. /ID# 142793, Monroe, Louisiana
  - Vanguard Medical Research, LLC /ID# 153123, Shreveport, Louisiana
  - MMP Women's Health /ID# 145612, Portland, Maine
  - The Center for Rheumatology & /ID# 142742, Wheaton, Maryland
  - Mansfield Health Center /ID# 147628, Mansfield, Massachusetts
  - Clinical Pharmacology Study Gr /ID# 142744, Worcester, Massachusetts
  - June DO, PC /ID# 142756, Lansing, Michigan
  - North Mississippi Med Clinics /ID# 142781, Tupelo, Mississippi
  - Clayton Medical Associates dba Saint Louis Rheumatology /ID# 142745, St Louis, Missouri
  - Barbara Caciolo, MD /ID# 142749, St Louis, Missouri
  - Westroads Clinical Research /ID# 142802, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 145958, Lebanon, New Hampshire
  - Atlantic Coast Research /ID# 148347, Toms River, New Jersey
  - Ocean Rheumatology, PA /ID# 142785, Toms River, New Jersey
  - The Center for Rheumatology /ID# 142784, Albany, New York
  - North Shore University Hospital /ID# 142772, New Hyde Park, New York
  - Buffalo Rheumatology /ID# 142766, Orchard Park, New York
  - Joint & Muscle Research Instit /ID# 142797, Charlotte, North Carolina
  - DJL Clinical Research, PLLC /ID# 142769, Charlotte, North Carolina
  - Cape Fear Arthritis Care /ID# 148344, Leland, North Carolina
  - Coastal Carolina Health Care /ID# 148351, New Bern, North Carolina
  - Shanahan Rheuma & Immuno /ID# 142812, Raleigh, North Carolina
  - Trinity Health Med Arts Clinic /ID# 142754, Minot, North Dakota
  - Cincinnati Rheumatic Disease Study Group, Inc. /ID# 142791, Cincinnati, Ohio
  - STAT Research, Inc. /ID# 142821, Vandalia, Ohio
  - Health Research Oklahoma /ID# 142751, Oklahoma City, Oklahoma
  - Healthcare Research Consultant /ID# 142815, Tulsa, Oklahoma
  - East Penn Rheumatology Assoc /ID# 142790, Bethlehem, Pennsylvania
  - Clinical Research Ctr Reading /ID# 151714, Wyomissing, Pennsylvania
  - Columbia Arthritis Center /ID# 153728, Columbia, South Carolina
  - West Tennessee Research Inst /ID# 142739, Jackson, Tennessee
  - Arthritis Associates, PLLC /ID# 142774, Kingsport, Tennessee
  - Arthritis Associates, PLLC /ID# 155462, Kingsport, Tennessee
  - Dr. Ramesh Gupta /ID# 142767, Memphis, Tennessee
  - Tekton Research, Inc. /ID# 142805, Austin, Texas
  - Diagnostic Group Integrated He /ID# 148340, Beaumont, Texas
  - Arth and Osteo Clin Brazo Valley /ID# 148343, College Station, Texas
  - Arthritis Care and Diagnostic /ID# 151344, Dallas, Texas
  - Metroplex Clinical Research /ID# 142758, Dallas, Texas
  - Rheumatic Disease Clin Res Ctr /ID# 150914, Houston, Texas
  - Baylor College of Medicine /ID# 142753, Houston, Texas
  - Rheumatology Clinic of Houston /ID# 150915, Houston, Texas
  - Houston Institute for Clin Res /ID# 142768, Houston, Texas
  - Pioneer Research Solutions, Inc. /ID# 151346, Houston, Texas
  - Arthritis & Osteoporosis Assoc /ID# 147567, Lubbock, Texas
  - P&I Clinical Research /ID# 151345, Lufkin, Texas
  - SW Rheumatology Res. LLC /ID# 142813, Mesquite, Texas
  - Trinity Universal Research Association /ID# 149278, Plano, Texas
  - Arthritis & Osteo Ctr of S. TX /ID# 142773, San Antonio, Texas
  - Arthritis Clinic of Central TX /ID# 148346, San Marcos, Texas
  - DM Clinical Research /ID# 151007, Tomball, Texas
  - Arthritis & Osteoporosis Clinic /ID# 142760, Waco, Texas
  - Western Washington Arthritis C /ID# 142776, Bothell, Washington
  - Arthritis Northwest, PLLC /ID# 150924, Spokane, Washington
  - The Vancouver Clinic, INC. PS /ID# 147946, Vancouver, Washington
  - West Virginia Research Inst /ID# 153087, South Charleston, West Virginia
  - Aurora Rheumatology and Immunotherapy Center /ID# 142820, Franklin, Wisconsin
- Australia (2):
  - The Queen Elizabeth Hospital /ID# 142419, Woodville, South Australia
  - Emeritus Research /ID# 142416, Camberwell, Victoria
- Austria (5):
  - Medizinische Universität Wien /ID# 142424, Vienna, Vienna
  - Universitaetsklinik fuer Inner /ID# 142423, Graz
  - Rheuma Zentrum Favoriten GmbH /ID# 142421, Vienna
  - Rheuma-Zentrum Wien-Oberlaa /ID# 142425, Vienna
  - Wilhelminenspital der Stadt Wien /ID# 142422, Vienna
- Belgium (5):
  - Cliniques Universitaires Saint Luc /ID# 142426, Woluwe-Saint-Lambert, Brussels Capital
  - Rhumaconsult SPRL /ID# 151378, Charleroi, Hainaut
  - UZ Gent /ID# 142429, Ghent, Oost-Vlaanderen
  - ReumaClinic Genk /ID# 142431, Genk
  - AZ Damiaan /ID# 142427, Ostend
- Ciads /Id# 142526, Winnipeg, Manitoba, Canada
- Czechia (2):
  - Revmatologie MUDr. Klara Sirova /ID# 142536, Ostrava
  - Medical Plus, s.r.o. /ID# 148345, Uherské Hradište
- Estonia (2):
  - MediTrials /ID# 151777, Tartu, Tartu
  - East Tallinn Central Hospital /ID# 142543, Tallinn
- Finland (2):
  - Kiljava Medical Research /ID# 142546, Hyvinkää
  - Paijat-Hame Central Hospital /ID# 149185, Lahti
- France (7):
  - CHR Orleans - Hopital de la Source /ID# 142557, Orléans, Centre-Val de Loire
  - Hopital Universitaire Purpan /ID# 144697, Toulouse, Haute-Garonne
  - Hopital Saint Eloi /ID# 142552, Montpellier, Herault
  - Centre Hospitalier Le Mans /ID# 145956, Le Mans, Sarthe
  - CHU Bordeaux-Hopital Pellegrin /ID# 144700, Bordeaux
  - Centre Hospitalier Jean Rougie /ID# 142556, Cahors
  - Hopital Edouard Herriot /ID# 144698, Lyon
- Germany (9):
  - Uniklinik Koln /ID# 142563, Cologne, North Rhine-Westphalia
  - Rheumazentrum Ruhrgebiet /ID# 145600, Herne, North Rhine-Westphalia
  - Charité Universitätsmedizin Campus Mitte /ID# 142559, Berlin
  - Rheumaforschungszentrum II /ID# 142560, Hamburg
  - Schoen Klinikum Hamburg Eilbek /ID# 142566, Hamburg
  - Asklepios Klinik Altona /ID# 142561, Hamburg
  - LMU Klinikum der Universität München /ID# 142564, Munich
  - MVZ Planegg /ID# 142565, Planegg
  - Knappschaftsklinikum Saar /ID# 142562, Püttlingen
- General Hospital of Athens Laiko /ID# 142579, Athens, Attica, Greece
- Hungary (4):
  - Vital Medical Center Orvosi es /ID# 142586, Veszprém, Veszprém megye
  - Revita Reumatologiai Rendelo /ID# 142590, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 142587, Debrecen
  - Bekes Megyei Pandy Kalman Korh /ID# 142588, Gyula
- St Vincent's University Hosp /ID# 142593, Dublin, Ireland
- Israel (3):
  - Tel Aviv Sourasky Medical Ctr /ID# 142597, Tel Aviv, Tel Aviv
  - Bnai Zion Medical Center /ID# 151945, Haifa
  - The Lady Davis Carmel MC /ID# 142599, Haifa
- Latvia (3):
  - LTD M+M Centers /ID# 142624, Ādaži
  - P. Stradins Clinical Univ Hosp /ID# 142623, Riga
  - Arthritis Clinic Ltd /ID# 153560, Riga
- Timaru Medical Specialists Ltd /ID# 142657, Timaru, New Zealand
- Poland (5):
  - Pratia MCM Krakow /ID# 142664, Krakow, Lesser Poland Voivodeship
  - WroMedica I. Bielicka, A. Strzalkowska s.c. /ID# 142665, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Pratia Warszawa /ID# 142667, Warsaw, Masovian Voivodeship
  - Centrum Medyczne AMED Warszawa Targowek /ID# 142663, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 142666, Gdynia, Pomeranian Voivodeship
- Portugal (2):
  - Centro Hospitalar De Vila Nova /ID# 142670, Vila Nova de Gaia, Porto District
  - Centro Hospitalar Lisboa Norte, EPE /ID# 142668, Lisbon
- GCM Medical Group /ID# 142671, San Juan, Puerto Rico
- Family Outpatient clinic#4,LLC /ID# 150910, Korolev, Moscow, Russia
- Slovakia (3):
  - ARTROMAC n.o. /ID# 142692, Košice
  - Nemocnica Kosice Saca, a.s. /ID# 142693, Košice
  - Narodny ustav reumatickych chorob Piestany /ID# 142691, Pieštany
- South Korea (3):
  - Hanyang University Seoul Hospi /ID# 150883, Seoul, Seongdong-gu
  - Inha University Hospital /ID# 150881, Incheon
  - Seoul National University Hospital /ID# 142622, Seoul
- Spain (6):
  - H. Un. Marques de Valdecilla /ID# 142706, Santander, Cantabria
  - Hospital Regional de Malaga /ID# 142707, Málaga, Malaga
  - Comple Hosp Univ de A Coruna /ID# 142708, A Coruña
  - Hospital Clin Univ San Carlos /ID# 142711, Madrid
  - Clinica Gaias /ID# 142709, Santiago de Compostela
  - Hospital Universitario La Fe /ID# 142716, Valencia
- Sweden (4):
  - Sahlgrenska University Hosp /ID# 142720, Gothenburg
  - Capio Movement Halmstad /ID# 148236, Halmstad
  - Orebro Universitetssjukhuset /ID# 142718, Örebro
  - Vastmanlands Sjukhus /ID# 142721, Västerås
- Switzerland (2):
  - Universitaetsspital Basel /ID# 145610, Basel
  - HFR Fribourg - Hopital Canton /ID# 142723, Fribourg
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty /ID# 142729, Ankara
  - Ankara Ataturk Training & Res /ID# 142727, Ankara
  - Ondokuz mayis University Facul /ID# 142728, Samsun
- United Kingdom (7):
  - Whipps Cross Univ Hospital /ID# 145957, London, London, City of
  - The Royal Free Hospital /ID# 142733, London, London, City of
  - Mid Essex Hospitals NHS Trust /ID# 148992, Chelmsford
  - Western General Hospital /ID# 142732, Edinburgh
  - West Suffolk Hospital /ID# 148993, Ipswich
  - Arrowe Park Hospital /ID# 148991, Metropolitan Borough of Wirral
  - Queen Alexandra Hospital /ID# 142735, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Genovese MC, Fleischmann R, Combe B, Hall S, Rubbert-Roth A, Zhang Y, Zhou Y, Mohamed MF, Meerwein S, Pangan AL. Safety and efficacy of upadacitinib in patients with active rheumatoid arthritis refractory to biologic disease-modifying anti-rheumatic drugs (SELECT-BEYOND): a double-blind, randomised controlled phase 3 trial. Lancet. 2018 Jun 23;391(10139):2513-2524. doi: 10.1016/S0140-6736(18)31116-4. Epub 2018 Jun 18. PMID 29908670
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] van Vollenhoven RF, Hall S, Wells AF, Meerwein S, Song Y, Tanjinatus O, Fleischmann R. Long-term sustainability of response to upadacitinib among patients with active rheumatoid arthritis refractory to biological treatments: results up to 5 years from SELECT-BEYOND. RMD Open. 2024 Jul 24;10(3):e004037. doi: 10.1136/rmdopen-2023-004037. PMID 39053948
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Fleischmann R, Curtis JR, Charles-Schoeman C, Mysler E, Yamaoka K, Richez C, Palac H, Dilley D, Liu J, Strengholt S, Burmester G. Safety profile of upadacitinib in patients at risk of cardiovascular disease: integrated post hoc analysis of the SELECT phase III rheumatoid arthritis clinical programme. Ann Rheum Dis. 2023 Sep;82(9):1130-1141. doi: 10.1136/ard-2023-223916. Epub 2023 Jun 12. PMID 37308218
- [Derived] Conaghan PG, Pavelka K, Hsieh SC, Bonnington TL, Kent TC, Marchbank K, Edwards CJ. Evaluating the efficacy of upadacitinib in patients with moderate rheumatoid arthritis: a post-hoc analysis of the SELECT phase 3 trials. Rheumatol Adv Pract. 2023 Feb 8;7(1):rkad017. doi: 10.1093/rap/rkad017. eCollection 2023. PMID 36794283
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Kakehasi AM, Radominski SC, Baravalle MD, Palazuelos FCI, Garcia-Garcia C, Arruda MS, Curi M, Liu J, Qiao M, Velez-Sanchez P, Vargas JI. Safety of upadacitinib in Latin American patients with rheumatoid arthritis: an integrated safety analysis of the SELECT phase 3 clinical program. Clin Rheumatol. 2023 May;42(5):1249-1258. doi: 10.1007/s10067-023-06513-y. Epub 2023 Jan 30. PMID 36715850
- [Derived] Bergman M, Buch MH, Tanaka Y, Citera G, Bahlas S, Wong E, Song Y, Zueger P, Ali M, Strand V. Routine Assessment of Patient Index Data 3 (RAPID3) in Patients with Rheumatoid Arthritis Treated with Long-Term Upadacitinib Therapy in Five Randomized Controlled Trials. Rheumatol Ther. 2022 Dec;9(6):1517-1529. doi: 10.1007/s40744-022-00483-4. Epub 2022 Sep 20. PMID 36125701
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Cohen SB, van Vollenhoven RF, Winthrop KL, Zerbini CAF, Tanaka Y, Bessette L, Zhang Y, Khan N, Hendrickson B, Enejosa JV, Burmester GR. Safety profile of upadacitinib in rheumatoid arthritis: integrated analysis from the SELECT phase III clinical programme. Ann Rheum Dis. 2021 Mar;80(3):304-311. doi: 10.1136/annrheumdis-2020-218510. Epub 2020 Oct 28. PMID 33115760
- [Derived] Strand V, Schiff M, Tundia N, Friedman A, Meerwein S, Pangan A, Ganguli A, Fuldeore M, Song Y, Pope J. Effects of upadacitinib on patient-reported outcomes: results from SELECT-BEYOND, a phase 3 randomized trial in patients with rheumatoid arthritis and inadequate responses to biologic disease-modifying antirheumatic drugs. Arthritis Res Ther. 2019 Dec 2;21(1):263. doi: 10.1186/s13075-019-2059-8. PMID 31791386
- [Derived] Nader A, Mohamed MF, Winzenborg I, Doelger E, Noertersheuser P, Pangan AL, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy and Safety in Phase II and III Studies to Support Benefit-Risk Assessment in Rheumatoid Arthritis. Clin Pharmacol Ther. 2020 Apr;107(4):994-1003. doi: 10.1002/cpt.1671. Epub 2019 Nov 30. PMID 31610021
- See also: Related Info. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 152 sites located in 26 countries from March 2016 to January 2017. Eligible participants had active rheumatoid arthritis (RA) and previous inadequate response or intolerance to biologic disease-modifying anti-rheumatic drugs (bDMARDs), and were receiving concomitant background conventional synthetic DMARDS (csDMARDs).
Pre-assignment Details: Participants were randomized in a 1:1:2:2 ratio to one of the four treatment groups below. Randomization was stratified by the number of previous bDMARDs used and geographic region.
Groups:
- Placebo / Upadacitinib 15 mg: Participants randomized to receive placebo once daily for 12 weeks followed by upadacitinib 15 mg once daily from Week 12 to Week 260.
- Placebo / Upadacitinib 30 mg: Participants randomized to receive placebo once daily for 12 weeks followed by upadacitinib 30 mg once daily from Week 12 to Week 260. After Protocol Amendment 4 participants still on study were switched to receive upadacitinib 15 mg.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily for 12 weeks followed by upadacitinib 15 mg once daily from Week 12 to Week 260.
- Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily for 12 weeks followed by upadacitinib 30 mg once daily from Week 12 to Week 260. After Protocol Amendment 4 participants still on study were switched to receive upadacitinib 15 mg.
Period: Period 1: Day 1 to Week 12
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 85 | 84 | 165 | 165
Received Study Treatment | 85 | 84 | 164 | 165
Completed | 75 | 76 | 157 | 149
Not Completed | 10 | 8 | 8 | 16
Not completed — Adverse Event | 2 | 2 | 1 | 12
Not completed — Withdrawal by Subject | 2 | 1 | 4 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Other | 4 | 4 | 2 | 2
Not completed — Randomized in Error | 0 | 0 | 1 | 0
Period: Period 1: Week 12 to Week 24
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 75 | 76 | 157 | 149
Received Study Treatment | 72 | 75 | 156 | 148
Completed | 72 | 74 | 153 | 135
Not Completed | 3 | 2 | 4 | 14
Not completed — Adverse Event | 1 | 2 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 1 | 4
Period: Period 2: Week 24 to Week 260
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started (Six participants completed the Week 24 visit but did not continue into Period 2.) | 71 | 73 | 152 | 132
Switched to Upadacitinib 15 mg After Protocol Amendment 4 | 0 | 44 | 0 | 94
Completed | 35 | 41 | 81 | 82
Not Completed | 36 | 32 | 71 | 50
Not completed — Adverse Event | 11 | 9 | 21 | 11
Not completed — Withdrawal by Subject | 11 | 10 | 17 | 10
Not completed — Lost to Follow-up | 1 | 5 | 9 | 6
Not completed — Lack of Efficacy | 5 | 3 | 9 | 8
Not completed — Other | 8 | 5 | 15 | 15

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug. The 2 placebo groups were combined for analysis of data through Week 12.
Groups:
- Placebo: Participants received placebo once daily for 12 weeks.
- Upadacitinib 15 mg: Participants received upadacitinib 15 mg once daily for 12 weeks.
- Upadacitinib 30 mg: Participants received upadacitinib 30 mg once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 169 | 164 | 165 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.39) | 56.3 (11.34) | 57.3 (11.55) | 57.1 (11.42)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 14 | 11 | 14 | 39
  40 - 64 years | 106 | 115 | 103 | 324
  ≥ 65 years | 49 | 38 | 48 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 137 | 138 | 418
  Male | 26 | 27 | 27 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 34 | 28 | 86
  Not Hispanic or Latino | 145 | 130 | 137 | 412
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 143 | 142 | 148 | 433
  Black or African American | 21 | 17 | 10 | 48
  American Indian/Alaska Native | 0 | 3 | 4 | 7
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 1
  Asian | 5 | 2 | 2 | 9
Geographic Region [Count of Participants; unit: Participants] — Other includes Australia, New Zealand, and Israel.
  Participants
    North America | 110 | 109 | 109 | 328
    Western Europe | 33 | 32 | 32 | 97
    Eastern Europe | 23 | 22 | 22 | 67
    Asia | 0 | 0 | 1 | 1
    Other | 3 | 1 | 1 | 5
Prior Failed Biological Disease-modifying Anti-rheumatic Drugs (bDMARDs) [Count of Participants; unit: Participants] — Randomization was stratified by the number of previous bDMARDs used:
  Stratum 1 consisted of participants who had inadequate response or intolerance to one or two biologics of the same class;
  Stratum 2 consisted of participants who had inadequate response or intolerance to at least three biologics of the same class and/or at least two biologics with different mechanisms of action.
  Participants
    Stratum 1 | 117 | 116 | 111 | 344
    Stratum 2 | 52 | 48 | 54 | 154
Duration of RA Diagnosis [Mean (Standard Deviation); unit: years] | 14.5 (9.22) | 12.4 (9.38) | 12.7 (9.65) | 13.2 (9.45)
Concomitant Conventional Synthetic DMARD Use at Baseline [Count of Participants; unit: Participants]
  Methotrexate alone | 122 | 118 | 124 | 364
  Methotrexate and other csDMARD | 17 | 19 | 11 | 47
  csDMARD other than methotrexate | 29 | 24 | 29 | 82
  Missing | 1 | 3 | 1 | 5
Tender Joint Count [Mean (Standard Deviation); unit: tender joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  tender joints | 28.5 (15.27) | 27.8 (16.31) | 27.3 (15.23) | 27.9 (15.58)
Swollen Joint Count [Mean (Standard Deviation); unit: swollen joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  swollen joints | 16.3 (9.58) | 17.0 (10.75) | 17.2 (11.37) | 16.8 (10.57)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: mm] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale (VAS) from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain." Population: Participants with available data
  mm
    number analyzed (Participants) | 166 | 163 | 161 | 490
    (all) | 68.9 (21.03) | 68.2 (19.77) | 65.3 (20.67) | 67.5 (20.52)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 166 | 163 | 163 | 492
    (all) | 66.3 (22.72) | 67.2 (19.60) | 64.7 (21.05) | 66.1 (21.15)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a VAS scale from 0 to 100 mm, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 161 | 157 | 157 | 475
    (all) | 66.9 (16.92) | 68.7 (16.59) | 66.4 (15.63) | 67.3 (16.39)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 166 | 163 | 161 | 490
    (all) | 1.6 (0.60) | 1.7 (0.64) | 1.6 (0.59) | 1.6 (0.61)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 16.3 (21.10) | 16.2 (18.62) | 16.0 (21.23) | 16.2 (20.32)
Disease Activity Score 28 Based on CRP (DAS28[CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28 score > 5.1 indicates high disease activity, a DAS28 score ≤ 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 166 | 163 | 163 | 492
    (all) | 5.8 (1.00) | 5.9 (0.95) | 5.8 (0.89) | 5.8 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: The primary endpoint for United States (US)/Food and Drug Administration (FDA) regulatory purposes was ACR 20% response (ACR20) at Week 12. Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 169 | 164 | 165
percentage of participants | 28.4 [21.6 to 35.2] | 64.6 [57.3 to 72.0] | 56.4 [48.8 to 63.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — The overall type I error rate of the primary and ranked key secondary endpoints for the two doses was controlled using a graphical multiple testing procedure; p < 0.001, Cochran-Mantel-Haenszel — The adjusted p-value under multiplicity control is reported, with significance achieved if the adjusted p-value is less than 0.05; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological DMARD use (stratum 1 vs stratum 2); Response Rate Difference = 36.2, 95% CI 2-sided [26.2 to 46.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 28.0, 95% CI 2-sided [17.8 to 38.1] — Response Rate Difference = Upadacitinib - Placebo

2. Primary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 12
Description: The primary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes was low disease activity, based on a Disease Activity Score 28 (DAS28)-CRP score of ≤ 3.2 at Week 12.
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score less than or equal to 3.2 indicates low disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 169 | 164 | 165
percentage of participants | 14.2 [8.9 to 19.5] | 43.3 [35.7 to 50.9] | 42.4 [34.9 to 50.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 29.1, 95% CI 2-sided [19.9 to 38.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 28.2, 95% CI 2-sided [19.0 to 37.4] — Response Rate Difference = Upadacitinib - Placebo

3. Secondary Outcome: Change From Baseline in in Disease Activity Score 28 (CRP) at Week 12
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data at baseline; multiple imputation was used for missing post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 165 | 163 | 161
units on a scale | -1.02 [-1.23 to -0.80] | -2.31 [-2.52 to -2.10] | -2.29 [-2.50 to -2.09]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of covariance (ANCOVA) model with treatment, prior biological DMARD use (stratum 1 vs stratum 2) and baseline value as covariates; LS Mean Difference = -1.29, 95% CI 2-sided [-1.57 to -1.01] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment, prior biological DMARD use (stratum 1 vs stratum 2) and baseline value as covariates; LS Mean Difference = -1.28, 95% CI 2-sided [-1.56 to -0.99] — Treatment Difference = Upadacitinib - Placebo

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data at baseline; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 165 | 163 | 160
units on a scale | -0.17 [-0.26 to -0.08] | -0.39 [-0.48 to -0.30] | -0.42 [-0.51 to -0.33]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment, prior biological DMARD use (stratum 1 vs stratum 2) and baseline value as covariates; LS Mean Difference = -0.22, 95% CI 2-sided [-0.34 to -0.10] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment, prior biological DMARD use (stratum 1 vs stratum 2) and baseline value as covariates; LS Mean Difference = -0.25, 95% CI 2-sided [-0.38 to -0.13] — Treatment Difference = Upadacitinib - Placebo

5. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 145 | 156 | 147
units on a scale | 2.39 [1.14 to 3.64] | 5.83 [4.60 to 7.05] | 7.02 [5.78 to 8.25]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; MMRM model with fixed effects of treatment, visit, and treatment-by-visit interaction, previous bDMARD use, and baseline value as covariate; LS Mean DIfference = 3.44, 95% CI 2-sided [1.72 to 5.15] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 4.63, 95% CI 2-sided [2.89 to 6.36] — Treatment Difference = Upadacitinib - Placebo

6. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 169 | 164 | 165
percentage of participants | 11.8 [7.0 to 16.7] | 34.1 [26.9 to 41.4] | 35.8 [28.4 to 43.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 22.3, 95% CI 2-sided [13.6 to 31.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 23.9, 95% CI 2-sided [15.1 to 32.7] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 169 | 164 | 165
percentage of participants | 6.5 [2.8 to 10.2] | 11.6 [6.7 to 16.5] | 23.0 [16.6 to 29.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p = 0.110, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 5.1, 95% CI 2-sided [-1.1 to 11.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 16.5, 95% CI 2-sided [9.1 to 23.9] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 1
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and week 1
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 1 or for whom ACR data were missing at Week 1 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 169 | 164 | 165
percentage of participants | 10.7 [6.0 to 15.3] | 27.4 [20.6 to 34.3] | 24.8 [18.3 to 31.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 16.8, 95% CI 2-sided [8.5 to 25.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 14.2, 95% CI 2-sided [6.1 to 22.3] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: Adverse events are reported for Weeks 1 to 12 (all participants) and from Weeks 1 to 260 for participants who received upadacitinib.
Groups:
- Placebo: Weeks 1-12: Participants received placebo once daily for 12 weeks.
- Upadacitinib 15 mg: Weeks 1-12: Participants received upadacitinib 15 mg once daily for 12 weeks.
- Upadacitinib 30 mg: Weeks 1-12: Participants received upadacitinib 30 mg once daily for 12 weeks.
- Upadacitinib 15 mg: Weeks 1-260: Participants originally randomized to upadacitinib 15 mg received upadacitinib 15 mg for 260 weeks and participants originally randomized to placebo followed by upadacitinib 15 mg received upadacitinib 15 mg from Week 12 to Week 260.
- Upadacitinib 30 mg: Weeks 1-260/Switch: Participants originally randomized to upadacitinib 30 mg received upadacitinib 30 mg up to implementation of Protocol Amendment 4 (December 2019) and participants originally randomized to placebo followed by upadacitinib 30 mg received upadacitinib 30 mg from Week 12 up to Week 260 or implementation of Protocol Amendment 4.
- Upadacitinib 15 mg After Switch: Participants who were receiving upadacitinib 30 mg in Period 2 were switched to upadacitinib 15 mg once daily after implementation of Protocol Amendment 4 (December 2019) up to Week 260.
Arm/Group | Placebo: Weeks 1-12 | Upadacitinib 15 mg: Weeks 1-12 | Upadacitinib 30 mg: Weeks 1-12 | Upadacitinib 15 mg: Weeks 1-260 | Upadacitinib 30 mg: Weeks 1-260/Switch | Upadacitinib 15 mg After Switch
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/164 | 1/165 | 9/236 | 5/240 | 2/138
Serious Adverse Events (participants affected / at risk) | 0/169 | 9/164 | 12/165 | 87/236 | 71/240 | 21/138
Other Adverse Events (participants affected / at risk) | 68/169 | 68/164 | 78/165 | 196/236 | 203/240 | 59/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: Weeks 1-12 (N=169) | Upadacitinib 15 mg: Weeks 1-12 (N=164) | Upadacitinib 30 mg: Weeks 1-12 (N=165) | Upadacitinib 15 mg: Weeks 1-260 (N=236) | Upadacitinib 30 mg: Weeks 1-260/Switch (N=240) | Upadacitinib 15 mg After Switch (N=138)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid cyst (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Volvulus of small bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Cavernous sinus thrombosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perinephric abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 9 (10) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis aspergillus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 7 (9) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device material issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device pacing issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (8) | 3 (4) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (2) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
May-Thurner syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: Weeks 1-12 (N=169) | Upadacitinib 15 mg: Weeks 1-12 (N=164) | Upadacitinib 30 mg: Weeks 1-12 (N=165) | Upadacitinib 15 mg: Weeks 1-260 (N=236) | Upadacitinib 30 mg: Weeks 1-260/Switch (N=240) | Upadacitinib 15 mg After Switch (N=138)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 12 (12) | 11 (13) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4) | 5 (7) | 13 (14) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 15 (16) | 9 (9) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (5) | 5 (7) | 12 (14) | 23 (25) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 7 (7) | 14 (15) | 19 (23) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5) | 5 (5) | 14 (17) | 11 (12) | 0 (0)
Fatigue (General disorders) | 3 (4) | 0 (0) | 7 (7) | 4 (5) | 16 (16) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 11 (11) | 14 (15) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 2 (2) | 13 (16) | 7 (9) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 7 (7) | 4 (4) | 27 (32) | 37 (41) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 2 (2) | 7 (7)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 12 (13) | 15 (20) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 22 (25) | 32 (38) | 8 (9)
Nasopharyngitis (Infections and infestations) | 11 (11) | 7 (8) | 9 (9) | 34 (67) | 41 (56) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 13 (15) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 14 (14) | 11 (11) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 22 (34) | 19 (24) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 13 (14) | 11 (11) | 74 (116) | 67 (116) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (11) | 16 (19) | 9 (10) | 43 (77) | 49 (79) | 11 (13)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (2) | 4 (4) | 14 (17) | 18 (24) | 7 (7)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 18 (21) | 27 (33) | 4 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 13 (13) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 15 (16) | 7 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 2 (4) | 26 (34) | 28 (37) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 16 (19) | 15 (17) | 8 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (9) | 13 (14) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 14 (15) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 13 (16) | 8 (8) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (5) | 6 (6) | 34 (53) | 39 (51) | 13 (17)
Headache (Nervous system disorders) | 9 (9) | 7 (7) | 8 (8) | 17 (19) | 19 (23) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4) | 9 (9) | 13 (13) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1) | 8 (8) | 13 (14) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) | 28 (36) | 19 (20) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 2 (2) | 13 (13) | 8 (9) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 13 (13) | 16 (20) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 3 (3) | 29 (32) | 19 (22) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT02706847/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT02706847/SAP_003.pdf